CLINICAL TRIAL: NCT00759421
Title: An Exploratory Cognition Study Conducted as an add-on to Clinical Trial 11286, to Evaluate the Neurocognitive Effects of 12 Weeks Treatment With Sertindole and Olanzapine in Patients With Schizophrenia
Brief Title: Exploratory Cognition Study of Sertindole in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11286B
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — sertindole; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Sertindole
- 2 (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Sertindole — 12 to 20 mg daily after initial up-titration, encapsulated tablets, orally, 84 days
  Arms: 1
Drug: Olanzapine — 10 to 20 mg daily after initial up-titration, encapsulated tablets, orally, 84 days
  Other Names: Zyprexa
  Arms: 2

SUMMARY:
The purpose of this exploratory study is to evaluate the effects of sertindole and olanzapine on neurocognitive functioning in patients with schizophrenia.

DETAILED DESCRIPTION:
Cognitive deficits, including impairments in areas such as memory, attention, and executive function, are major determinants and predictors of long-term disability in schizophrenia. At present, available antipsychotic medications are relatively ineffective in improving cognition. However, scientific discoveries during the past decade suggest that it may be possible to develop medications that are effective in improving cognition in schizophrenia.

One of the important reasons to focus on cognitive deficits as a target for pharmacological treatment, is the association found between cognitive impairment and social dysfunction observed in patients with schizophrenia. Pervasive cognitive deficits have a limiting effect on the quality of life of patients with schizophrenia including social interaction and problem solving, community living, and employment prospects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia
* Participation in 11286 study
* Capable of completing all study-related psychometric activities for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Global cognitive composite score | 12 weeks

SECONDARY OUTCOMES:
Cognitive performance in the following domains: 1) Working memory; 2) Attention and vigilance; 3) Verbal learning and memory; 4) Visual learning and memory; 5) Reasoning and problem solving; 6) Speed of processing | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- TWN001, Tapei, Taiwan